CLINICAL TRIAL: NCT04711980
Title: Efficacy and Safety of Mudan Granule (Combined With Methylcobalamin) on Type 2 Diabetic Peripheral Neuropathy: A Randomized,Double-blind,Placebo-controlled, Parallel-arm,Multi-center Trial
Brief Title: Post-marketing Evaluation of Mudan Granule Intervention on Type 2 Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fengmei Lian (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); The Affiliated Hospital of Qingdao University (Other); Chengdu University of Traditional Chinese Medicine (Other); The Fourth People's Hospital of Chongqing (Unknown); Zhengzhou Yihe Hospital Affiliated to Henan University (Unknown); Zhu Xianyi Memorial Hospital of Tianjin Medical University (Unknown); The Third Hospital of Xi'an (Unknown); Huashan Hospital (Other); Gansu Provincial People's Hospital (Unknown); Shenzhen Hospital of Guangzhou University of Traditional Chinese Medicine (Unknown); Affiliated Hospital of Changchun University of Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Fengmei Lian, chief physician, Professor, endocrinology department of Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020 Mudan Granule
Record Dates: First submitted 2021-01-07; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Peripheral Neuropathy Type 2
Keywords: Type 2 Diabetes Mellitus; diabetic peripheral neuropathy; Mudan granule
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mudan granule (Experimental): Based on the standard medical care, experimental group were treated with Mudan Granule 7g , 3 times/d.
  Intervention: Drug: Mudan granule
  Interventions: Drug: Mudan granule
- Placebo (Placebo Comparator): Based on the standard medical care, placebo-controlled group were treated with Placebo 7g , 3 times/d Intervention: Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mudan granule — Mudan granule,a traditional Chinese medicine formula,consists of nine Chinese herbs.
  Other: Standard medical care.Standard medical care is in accordance with China Guideline for type 2 diabetes (2013).
  Other Names: Mudan particle
  Arms: Mudan granule
Drug: Placebo — Granule(Placebo) is in accordance with Mudan granule in appearance, colour, taste.
  Other: Standard medical care. Standard medical care is in accordance with China Guideline for type 2 diabetes (2013).
  Other Names: Placebos
  Arms: Placebo

SUMMARY:
Background: Diabetic peripheral neuropathy (DPN) is a common and disabling chronic microvascular complications in patients with type 2 diabetic Mellitus (T2DM) that is characterized by nerve damage, affecting at least half of patients diagnosed with diabetes. It has been reported that DPN significantly contributes to the increased morbidity with diabetic foot ulcers by 60% and amputation by 85% that seriously threaten the quality of life. Mudan granule, a traditional Chinese medicinal preparation, is widely used in clinical practice for DPN in China. Evidence from clinical and preclinical studies have shown that Mudan granule could relieve symptoms and reduce the incidence of DPN exacerbations. However, the previous studies are of variable quality and poorly standardized,which limits the clinical application of Mudan granule. This study evaluates the efficacy and safety of Mudan granule combined with methylcobalamin in the treatment of type 2 diabetic peripheral neuropathy, providing the highest level of evidence of Mudan granule.

Methods and design: A randomized, double-blind, placebo-controlled,parallel-arm, and multi-centric clinical trial design was used based on a co-regimen of methylcobalamin. Subjects who met the inclusion criteria were randomly divided into two groups. The patients in the study group were treated with Mudan granule combined with methylcobalamin, and the patients in the control group were treated with placebo combined with methylcobalamin. The total intervention period is 24 weeks. The sample size was 402 cases.

Major evaluation indicators: Michigan Diabetic Neuropathy Score (MDNS) changes, the changes of MDNS were compared between the two groups before and after medication, adopting the evaluation method of difference values. Secondary Evaluation Indicators:(1) nerve conduction velocity changes, the changes in nerve conduction velocity of each nerve were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. (2)corneal nerve fiber density changes, the changes in corneal nerve fiber density of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. (3)corneal nerve branch density changes, the changes in corneal nerve branch density of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. (4)corneal nerve fiber length changes, the changes in corneal nerve fiber length of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. (5)Toronto Clinical Scoring System (TCSS) changes, the changes of toronto clinical score were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. (6)Traditional Chinese Medicine(TCM) syndromes efficacy score changes, the changes in TCM syndromes efficacy score were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. (7) Clinical symptoms score changes, the changes of each of clinical symptoms score were compared between the two groups before and after medication, adopting the evaluation method of difference values.

Discussion: We postulate that patients with type 2 diabetic peripheral neuropathy will benefit from therapy with Mudan granule.

DETAILED DESCRIPTION:
1. Research objective: To evaluate the efficacy and safety of Mudan granule combined with methylcobalamin in the treatment of type 2 diabetic peripheral neuropathy, providing the highest level of evidence of Mudan granule.
2. Experimental Measures and contrast: A randomized, double-blind, placebo-controlled,parallel- arm,and multi-centric clinical trial design was used on the basis of a co-regimen of methylcobalamin.The patients in the study group were treated with Mudan granule (7g 3 times/day for 24 weeks)and patients were treated with placebo (7g 3 times/day for 24 weeks) in the control group.The sample size was determined to 402 cases through statistics calculation.

   Sample size calculation basis: According to the previous study of Mudan granule combined with methylcobalamin in the treatment of DPN with 12 weeks intervention, the results of the MDNS indicated that the study group (Mudan granule + methylcobalamin) scale score was 5.48±1.19, and the control group (placebo + methylcobalamin) scale score was 8.21 ±1.24, and the mean difference between the two groups was 2.73;Assuming that Mudan granule combined with methylcobalamin in the treatment of DPN can reduce the MDNS by 0.58 after 12 weeks of intervention, it is considered better than the control group.Taking α=0.05, β=0.10, the study group and the control group with 24 weeks intervention were allocated at a ratio of 1:1. The sample size calculated by the Power Analysis and Sample Size (PASS) 11 software was not less than 167 cases in each group. Considering no more than 20% withdrawal rate, the total number of cases is 402, 201cases in each group.
3. Research design 3.1 This trial was designed as a randomized, double-blind, placebo-controlled,parallel-arm, and multi-centric clinical trial. Subjects who met the inclusion criteria were randomly divided into two groups. The patients in the study group were treated with Mudan granule combined with methylcobalamin , and the patients in the control group were treated with placebo combined with methylcobalamin. The sample size was 402 cases.

3.2 The total intervention period is 24 weeks. 3.3 Curative effect evaluation criteria 3.3.1 Major evaluation indicators Changes in total score on the Michigan Diabetic Neuropathy Score (MDNS) of Scale,MDNS was recorded on the Michigan Diabetic Neuropathy Score of Scale. The changes of MDNS were compared between the two groups before and after medication, adopting the evaluation method of difference values. The total score was 46, ranging from 0 (least severe) to 46 (most severe).

3.3.2 Secondary Evaluation Indicators

1. Changes in nerve conduction velocity,the changes in nerve conduction velocity of each nerve were compared between the two groups before and after taking medicine,adopting the evaluation method of difference values.
2. Changes in corneal nerve fiber density of each mm2,the changes in corneal nerve fiber density of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values.
3. Changes in corneal nerve branch density of each mm2,the changes in corneal nerve branch density of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values.
4. Changes in corneal nerve fiber length of each mm2,the changes in corneal nerve fiber length of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values.
5. Changes in total score on the Toronto Clinical Scoring System (TCSS) of Scale,toronto clinical score was recorded on the Toronto Clinical Scoring System(TCSS) of Scale. The changes of toronto clinical score were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. The total score was 19, ranging from 0 (least severe) to 19 (most severe).
6. Evaluation criteria of Traditional Chinese Medicine(TCM) syndromes efficacy score

   ①Clinical cure:TCM syndrome efficacy score reduced ≥90%.②Markedly effective: 90%>TCM syndrome efficacy score ≥70%.③Valid: 30% ≤ TCM syndrome efficacy score < 70%.④Invalid: TCM syndrome efficacy score reduced <30%.
7. Evaluation criteria of clinical symptoms score ①Disappearance: the symptoms disappeared,and the score was 0.②Improvement: the symptoms were relieved,and the score was reduced but not 0.③No improvement: the symptoms remained unchanged, and the score did not change.④Exacerbation: the symptoms exacerbated and the score increased.

3.4 Observation indicators

1. Demographic and clinical data:gender, age, disease course, family history,past medical history and so on (0 week).
2. Curative effect indicators：Michigan Diabetic Neuropathy Score (MDNS) (0,12,24weeks),nerve conduction velocity (0 weeks, 24 weeks),corneal nerve fiber parameters (0,24 weeks),Toronto Clinical Scoring System (TCSS) (0,12,24 weeks),TCM syndromes efficacy (0,4,8,12,16,20,24 weeks).
3. Monitoring indicators

   * Fasting blood glucose, blood pressure (0,4,8,12,16,20,24 weeks).

     * Glycated hemoglobin, blood lipid (0, 12, 24 weeks).
4. Safety indicators

   ①Adverse events (recorded in detail at any time).

   ②General vital signs:body temperature, heart rate, respiration and so on(0, 4, 8, 12, 16, 20, 24 weeks).

   ③Blood routine, urine routine, urine pregnancy test, stool routine, 12-lead Electrocardiography, liver and kidney function test (0, 12, 24 weeks).

   3.5 Basic treatment
   * Diabetes education.

     * Diabetic diet. ③Rational control of blood glucose: using oral hypoglycemic agents or insulin injections to keep all patients' blood glucose stable in the study. In principle, the type and dose of hypoglycemic agents should maintain unchanged. If fasting blood glucose fluctuates more than 20%,diabetes experts need to find and eliminate the predisposing factors as soon as possible, adjust the dose and monitor the blood glucose changes, so as to keep the blood glucose stable within 4 weeks.Adjusted dose of the drug needs to be detailed recorded in the combined medication table.

       * Taking methylcobalamin tablets (0.5mg,3 times/d). (Eisai (China) Pharmaceutical Co., Ltd.).

   3.6 Provisions for combined treatment

   ①All Chinese herbal medicines with the same efficacy as the study drug (including Chinese herbal medicines with similar therapeutic indications and Chinese herbal medicines with similar efficacy) were banned during the study period.

   ②Besides methylcobalamin, drugs such as alpha lipoic acid, epalrestat, and VitB12 for the treatment of diabetic peripheral neuropathy are prohibited.

   ③All combination therapy and treatment (treatment measure or treatment medicine of other diseases) should be documented in the combined medication table.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of type 2 diabetic peripheral neuropathy.
2. Meet the diagnostic criteria of TCM syndrome differentiation of qi deficiency and collaterals obstruction.
3. The patient's age is between 30-70 years.
4. At least 2 nerve conduction velocities have decreased on electromyography.
5. Sign informed consent.

Exclusion Criteria:

1. Recent use of antioxidants such as vitamin E or vitamin C, acute infection, liver and kidney dysfunction, acute complications of diabetes, severe cardiovascular and cerebrovascular diseases,neuropathy caused by long-term alcohol consumption and other factors.
2. Besides methylcobalamin,the drugs such as alpha lipoic acid, epalrestat, VitB12, Chinese patent medicine and decoction have been used to treat diabetic peripheral neuropathy within 4 weeks before enrollment.
3. Systolic blood pressure > 160 millimeters of mercury (mmHg) or diastolic blood pressure > 100mmHg.
4. Having the diabetic ketoacidosis, ketoacidosis and severe infection within one month.
5. Combined with cardiovascular, liver, kidney and hematopoietic system and other serious primary disease, serum transaminase beyond the normal value more than 2 times, serum creatinine greater than the upper limit of normal, psychiatric patients.
6. Pregnancy, prepared to pregnant or lactating women.
7. Having a history of multiple drug allergies or being allergic to the ingredients of Mudan granule.
8. Participate in other clinical studies within one month.
9. Drinking alcohol excessive and/or taking psychoactive substances, drug abusers and dependents over the past five years.
10. Having a history of active ophthalmopathy,ocular surgery,glaucoma,acute and chronic corneal diseases,extended-wearing contact lens and so on.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Changes in total score on the Michigan Diabetic Neuropathy Score (MDNS) of Scale | 0,12,24 weeks
  MDNS was recorded on the Michigan Diabetic Neuropathy Score of Scale. The changes of MDNS were compared between the two groups before and after medication, adopting the evaluation method of difference values. The total score was 46, ranging from 0 (least severe) to 46 (most severe).

SECONDARY OUTCOMES:
Changes in nerve conduction velocity | (0,24 weeks)
  The changes in nerve conduction velocity of each nerve were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values.
Changes in corneal nerve fiber density of each mm2 | (0,24 weeks)
  The changes in corneal nerve fiber density of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values.
Changes in corneal nerve branch density of each mm2 | (0,24 weeks)
  The changes in corneal nerve branch density of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values.
Changes in corneal nerve fiber length of each mm2 | (0,24 weeks)
  The changes in corneal nerve fiber length of each mm2 were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values.
Changes in total score on the Toronto Clinical Scoring System (TCSS) of Scale | (0,12,24 weeks)
  Toronto clinical score was recorded on the Toronto Clinical Scoring System(TCSS) of Scale. The changes of toronto clinical score were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. The total score was 19, ranging from 0 (least severe) to 19 (most severe).
Changes in total score on the Traditional Chinese Medicine(TCM) Syndromes Efficacy Score of Scale | (0,4,8,12,16,20,24 weeks)
  TCM syndromes efficacy score was recorded on the Traditional Chinese Medicine Syndromes Efficacy Score of Scale. The changes in TCM syndromes efficacy score were compared between the two groups before and after taking medicine, adopting the evaluation method of difference values. TCM syndromes efficacy score was 33, ranging from 0 (least severe) to 33 (most severe).
Changes in total score on the Clinical Symptoms Score of Scale | (0,12 ,24 weeks)
  Clinical symptoms score was recorded on the Clinical Symptoms Score of Scale.The changes of each of clinical symptoms score were compared between the two groups before and after medication,adopting the evaluation method of difference values. Each of clinical symptoms score was 6,ranging from 0 (least severe) to 6 (most severe). Clinical symptoms mainly included pain,numbness,paresthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Xin hua Xiao, Ph.D., Principal Investigator — Peking Union Medical College Hospital; Yi Li, Ph.D., Principal Investigator — Beijing Hospital; Shi jia Yu, Ph.D., Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; Yan gang Wang, Ph.D., Principal Investigator — The Affiliated Hospital of Qingdao University; Qiu Chen, Ph.D., Principal Investigator — Chengdu University of Traditional Chinese Medicine; Wu quan Deng, Ph.D., Principal Investigator — The Fourth People's Hospital of Chongqing; Zhi gang Zhao, Ph.D., Principal Investigator — Zhengzhou Yihe Hospital Affiliated to Henan University; Zhen qiang Song, Ph.D., Principal Investigator — Zhu Xianyi Memorial Hospital of Tianjin Medical University; Ping Liu, Master, Principal Investigator — The Third Hospital of Xi'an; Yi ming Li, Ph.D., Principal Investigator — Huashan Hospital; Jing Liu, Ph.D., Principal Investigator — Gansu Provincial People's Hospital; Chun Li Piao, Ph.D., Principal Investigator — Shenzhen Hospital of Guangzhou University of Traditional Chinese Medicine; Xiu ge Wang, Master, Principal Investigator — Affiliated Hospital of Changchun University of Chinese Medicine
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
Yes

REFERENCES:
- [Derived] Zhang Y, Jin D, Duan Y, Hao R, Chen K, Yu T, Lian F, Tong X. Efficacy of Mudan Granule (Combined With Methylcobalamin) on Type 2 Diabetic Peripheral Neuropathy: Study Protocol for a Double-Blind, Randomized, Placebo-Controlled, Parallel-Arm, Multi-Center Trial. Front Pharmacol. 2021 May 20;12:676503. doi: 10.3389/fphar.2021.676503. eCollection 2021. PMID 34093204